CLINICAL TRIAL: NCT03346122
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of JNJ-64991524 in Healthy Participants
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of JNJ-64991524 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108376; 2017-000229-11 (EudraCT Number); 64991524EDI1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1:JNJ-64991524 Dose Level (DL) 1 or Placebo(SAD Part 1) (Experimental): Participants will receive a single oral dose (Dose level 1) of either JNJ-64991524 or placebo capsules after an overnight fast (at least 10 hours) on Day 1 of Part 1.
  Interventions: Drug: JNJ-64991524 Dose Level 1; Drug: Placebo
- Cohort 2: JNJ-64991524 DL 2 or Placebo (SAD Part 1) (Experimental): Participants will receive a single oral dose (Dose level 2) of either JNJ-64991524 or placebo capsules after an overnight fast (at least 10 hours) on Day 1 of Part 1.
  Interventions: Drug: JNJ-64991524 Dose Level 2; Drug: Placebo
- Cohort 3: JNJ-64991524 DL 3 or Placebo (SAD Part 1) (Experimental): Participants will receive a single oral dose (Dose level 3) of either JNJ-64991524 or placebo capsules after an overnight fast (at least 10 hours) on Day 1 of Part 1.
  Interventions: Drug: JNJ-64991524 Dose Level 3; Drug: Placebo
- Cohort 4:JNJ-64991524 DL 4 or Placebo (SAD Part 1:Fasted-Fed) (Experimental): Participants will receive a single oral dose (Dose level 4) of either JNJ-64991524 or placebo capsules in a fasted condition on Day 1 and fed condition, on Day 7.
  Interventions: Drug: JNJ-64991524 Dose Level 4; Drug: Placebo
- Cohort 5: JNJ-64991524 DL 5 or Placebo (SAD Part 1) (Experimental): Participants will receive a single oral dose (Dose level 5) of JNJ-64991524 or placebo after an overnight fast (at least 10 hours) on Day 1 of Part 1.
  Interventions: Drug: JNJ-64991524 Dose Level 5; Drug: Placebo
- Cohort 6: JNJ-64991524 DL 6 or Placebo (SAD Part 1) (Experimental): Participants will receive a single oral dose (Dose level 6) of JNJ-64991524 or placebo after an overnight fast (at least 10 hours) on Day 1 of Part 1.
  Interventions: Drug: JNJ-64991524 Dose Level 6; Drug: Placebo
- Cohort 1: JNJ-64991524 DL 7 or Placebo (MAD Part 2) (Experimental): Participants will receive an oral dose (Dose level 7) JNJ-64991524 or placebo capsules once daily for 14 days in fasted or fed condition in Part 2. Fasted/fed condition will be determined based on tolerability and pharmacokinetics (PK) from Part 1.
  Interventions: Drug: Placebo; Drug: JNJ-64991524 Dose Level 7
- Cohort 2: JNJ-64991524 DL 8 or Placebo (MAD Part 2) (Experimental): Participants will receive an oral dose (Dose level 8) JNJ-64991524 or placebo capsules once daily for 14 days in fasted or fed condition in Part 2. Fasted/fed condition will be determined based on tolerability and PK from Part 1.
  Interventions: Drug: Placebo; Drug: JNJ-64991524 Dose Level 8
- Cohort 3: JNJ-64991524 DL 9 or Placebo (MAD Part 2) (Experimental): Participants will receive an oral dose (Dose level 9) JNJ-64991524 or placebo capsules once daily for 14 days in fasted or fed condition in Part 2. Fasted/fed condition will be determined based on tolerability and PK from Part 1.
  Interventions: Drug: Placebo; Drug: JNJ-64991524 Dose Level 9
- Cohort 4: JNJ-64991524 DL 6 or Placebo (MAD Part 2) (Experimental): Participants will receive an oral dose (Dose level 6) of JNJ-64991524 or placebo capsules once daily for 14 days in fasted or fed condition in Part 2. Fasted/fed condition will be determined by tolerability and PK from Part 1.
  Interventions: Drug: JNJ-64991524 Dose Level 6; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64991524 Dose Level 1 — Participants will receive JNJ-64991524 at a Dose Level 1 in SAD Part 1 of study.
  Arms: Cohort 1:JNJ-64991524 Dose Level (DL) 1 or Placebo(SAD Part 1)
Drug: JNJ-64991524 Dose Level 2 — Participants will receive JNJ-64991524 at a Dose Level 2 in SAD Part 1 of study.
  Arms: Cohort 2: JNJ-64991524 DL 2 or Placebo (SAD Part 1)
Drug: JNJ-64991524 Dose Level 3 — Participants will receive JNJ-64991524 at a Dose Level 3 in SAD Part 1 of study.
  Arms: Cohort 3: JNJ-64991524 DL 3 or Placebo (SAD Part 1)
Drug: JNJ-64991524 Dose Level 4 — Participants will receive JNJ-64991524 at a Dose Level 4 in SAD Part 1 of study.
  Arms: Cohort 4:JNJ-64991524 DL 4 or Placebo (SAD Part 1:Fasted-Fed)
Drug: JNJ-64991524 Dose Level 5 — Participants will receive JNJ-64991524 at a dose of Dose Level 5 in SAD Part 1 of study.
  Arms: Cohort 5: JNJ-64991524 DL 5 or Placebo (SAD Part 1)
Drug: JNJ-64991524 Dose Level 6 — Participants will receive JNJ-64991524 at a Dose Level 6 in SAD Part 1 and MAD part 2 of study.
  Arms: Cohort 4: JNJ-64991524 DL 6 or Placebo (MAD Part 2); Cohort 6: JNJ-64991524 DL 6 or Placebo (SAD Part 1)
Drug: Placebo — Participants will receive matching placebo in all cohorts on Day 1 in Part 1 and Part 2 of the study.
Drug: JNJ-64991524 Dose Level 7 — Participants will receive JNJ-64991524 at a dose of Dose Level 7 in MAD Part 2 of study for 14 days.
  Arms: Cohort 1: JNJ-64991524 DL 7 or Placebo (MAD Part 2)
Drug: JNJ-64991524 Dose Level 8 — Participants will receive JNJ-64991524 at a Dose Level 8 in MAD Part 2 of study for 14 days.
  Arms: Cohort 2: JNJ-64991524 DL 8 or Placebo (MAD Part 2)
Drug: JNJ-64991524 Dose Level 9 — Participants will receive JNJ-64991524 at a Dose Level 9 in MAD Part 2 of study for 14 days.
  Arms: Cohort 3: JNJ-64991524 DL 9 or Placebo (MAD Part 2)

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of JNJ-64991524 compared with placebo after administration of single ascending oral doses of JNJ-64991524 (Part 1) and multiple ascending oral doses of JNJ-64991524 (Part 2) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Weigh at least 50 kilogram (kg), and have a body mass index (BMI) of 18 kg/ meter (m)^2 to 30 kg/m^2, inclusive, at screening
* Be otherwise healthy on the basis of physical examination, medical history, vital signs, and 12-lead ECG performed at screening and Day-1. This determination must be recorded in the participant's source documents and initialed by the investigator
* Be otherwise healthy on the basis of clinical laboratory tests performed at screening and Day -1. If the results of the serum chemistry panel, including liver enzymes, white blood cell count and hematocrit, coagulation, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and confirmed initialed by the investigator
* Have the platelet count pretreatment clinical laboratory values not below the normal range during Screening and Day -1
* A woman must have a negative serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test on Day -2

Exclusion Criteria:

* History of liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Known allergies, hypersensitivity, or intolerance to JNJ-64991524 or its excipients
* History of severe allergic reaction, angioedema, or anaphylaxis to drugs or food
* Has a history of malignancy before screening. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or a malignancy which is considered cured with minimal risk of recurrence
* Has a history of or is infected with human immunodeficiency virus (HIV [positive serology for HIV antibody]); tests positive for hepatitis B virus (HBV) infection; has antibodies to hepatitis C virus (HCV) at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Part 1: Single Ascending Dose (SAD): Number of Participants with Treatment Emergent Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to Day 20
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Treatment-emergent were events between administration of study drug and up to Day 20 that were absent before treatment or that worsened relative to pre-treatment state.
Part 2: Multiple Ascending Dose (MAD): Number of Participants with Treatment Emergent Adverse Events as a Measure of Safety and Tolerability | Up to Day 28
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Treatment-emergent were events between administration of study drug and up to Day 28 that were absent before treatment or that worsened relative to pre-treatment state.
Number of Participants with Abnormalities in Vital Signs, Physical Examinations, Electrocardiogram (ECG), Cardiac Telemetry and Clinically Significant Laboratory Findings | Pre-dose, up to Day 20 (SAD) and up to Day 28 (MAD)
  Number of participants with abnormalities in vital signs, physical examinations, ECG, cardiac telemetry and clinically significant laboratory findings will be measured.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-64991524 | Pre-dose, up to Day 20 (SAD) and up to Day 28 (MAD)
  Plasma concentration assessment will be done to characterize the pharmacokinetics (PK) of JNJ-64991524.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Clinical Pharmacology Unit (located in ZNA Stuivenberg), Antwerp, Belgium